CLINICAL TRIAL: NCT01401517
Title: A Randomized, Double-blinded, Placebo-controlled, Phase IIa Dose-ranging Study to Assess the Safety, Pharmacokinetics, and Tolerability of Multiple Doses of Sodium Nitrite in Patients With Peripheral Arterial Disease (PAD) - SONIC
Brief Title: Phase IIa: Safety, PK, & Tolerability of Sodium Nitrite in Patients With Peripheral Arterial Disease-SONIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TheraVasc Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TheraVasc-TV1001-002
Record Dates: First submitted 2011-06-28; First posted 2011-07-25 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Microcrystalline cellulose NF at 60 mg/capsule, BID
  Interventions: Drug: sodium nitrite
- 40 mg Sodium Nitrite (Experimental): 40 mg dose, BID
  Interventions: Drug: sodium nitrite
- 80 mg Sodium Nitrite (Experimental): 80 mg dose, BID
  Interventions: Drug: sodium nitrite

INTERVENTIONS:
Drug: sodium nitrite — 0, 40 or 80 mg twice each day for 10 weeks followed by a 1 week escalation of 2 times the dose.
  Other Names: TV1001

SUMMARY:
Sodium nitrite has been demonstrated to promote new blood vessel growth, speed up wound healing and prevent tissue necrosis in animals. Since patients with PAD experience many of these problems, this study will seek to determine whether this drug, when given orally, could provide the same benefits to patients with PAD.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a manifestation of systemic atherosclerosis and a strong predictor of cardiovascular (CV) mortality. The systemic disease of atherosclerosis in these patients results in arterial stenoses in the arteries supplying the muscles of the lower extremities. During exercise, the stenoses limit the ability to increase blood flow, which leads to an oxygen supply/metabolic demand mismatch, a bio-energetic deficit, and subsequent muscle contractile dysfunction. Thus, the primary pathophysiology of PAD is related to the limitation in blood flow and abnormal hemodynamics (reduced tissue perfusion pressure and blood flow) of the lower limbs during exercise. Patients with PAD commonly present with symptoms of intermittent claudication (IC), often described by patients as a cramping, aching, or fatigue sensation in the calf muscles of the legs that occurs during physical activity. Notably, the symptom of claudication pain is due to exercise-induced ischemia in the muscles of the leg, causing a significant limitation of functional exercise capacity and adversely affecting quality of life.

Sodium nitrite is being investigated as a potential new therapy for improving function in patients with PAD. The overall goal of this dose-ranging study is to evaluate the safety, pharmacokinetics, tolerability, and potential biological activity of multiple doses of oral sodium nitrite in patients with PAD. As described above, the primary pathophysiology of PAD is related to the limitation in blood flow of the lower extremities, resulting in limited exercise tolerance and decreased quality of life. PAD is highly prevalent in patients with diabetes, leading to poor outcomes and accelerated disease progression compared with non-diabetic counter-parts. A common feature of both patient groups is endothelial dysfunction, decreased NO bioavailability, and depletion of NO stores, a finding that may be compounded when PAD and diabetic conditions coexist. Sodium nitrite is an inorganic salt that is found and metabolized in vivo. At physiological concentrations, sodium nitrite is known to cause vasodilation, a feature which is enhanced in hypoxic or ischemic environments. The nitrite anion acts a NO reservoir and can be readily converted to active NO by a non-enzymatic reaction with deoxyhemoglobin, making it a unique candidate for potential therapeutic effect in ischemic tissues. Accordingly, this study is designed to assess the safety and tolerability of sodium nitrite as well as the pharmacokinetic and pharmacodynamic relationship of sodium nitrite at two different doses versus placebo. Sodium nitrite's effects on endothelial function, a marker of NO bioactivity, and measures of functional walking capacity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between and including 35 and 85 years of age.
* Subjects must be either male or females post-menopausal, sterilized or using suitable birth control. Suitable birth control must be total abstinence, male partner sterilization or double barrier method paired with using oral contraception, injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, or intrauterine device (IUD).
* History of Peripheral Arterial Disease (PAD) confirmed by medical chart or an ankle brachial pressure index at rest ≤0.90.
* If receiving medical standard treatment for cardiac risk factors, subject must have been on a stable treatment for at least 1 month prior to Screening. Treatments must have not changed significantly in the last month and are not expected to change over the duration of the study.
* If subjects experience claudication symptoms, subjects must have stable lower extremity symptoms for at least 1 month prior to Screening.
* Ability to provide written informed consent and willingness as documented by a signed informed consent form.

Exclusion Criteria:

* Non-atherosclerotic PAD.
* Lower extremity surgical or percutaneous revascularization, evidence of graft failure or other peripheral vascular surgical procedure within last 6 months prior to Screening.
* Anticipated lower extremity revascularization within the treatment period.
* Myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack within 3 months prior to Screening.
* Poorly controlled diabetes (HgA1c > 10.0).
* Poorly controlled hypertension (systolic blood pressure (SBP) ≥ 160 mmHg or diastolic blood pressure (DBP) ≥ 100 mmHg) despite therapy.
* Systolic blood pressure ≤100 mmHg on current medical regimen.
* Hypersensitivity to sodium nitrite or related compounds.
* Renal insufficiency documented as eGFR < 30 mL/minute/1.73 m2.
* Pregnant or nursing women.
* Life expectancy < 6 months.
* A chronic illness that may increase the risks associated with this study in the opinion of the investigator.
* Active malignancy requiring active anti-neoplastic therapy that will, in the opinion of the investigator, interfere with study treatment or participation.
* Active infection.
* NYHA CHF Class III or IV.
* Recent hospitalization (< 30 days) for acute coronary syndrome, myocardial infarction, congestive heart failure or stroke.
* Recent (< 30 days) coronary revascularization.
* Previously treated with angiogenic factors or stem cell therapy within 1 year prior to Screening.
* Involvement in another PAD clinical trial within past 1 month prior to Screening.
* Exposed tendon, muscle or bone or a diagnosis of critical leg ischemia.
* Previous amputation within 3 months prior to Screening or planned amputation that would limit walking (e.g. small toe is allowed).
* The subject's ability to perform the 6 minute walk test is limited by symptoms other than claudication.
* Current diagnosis of alcohol or other substance abuse.
* History of methemoglobinemia, [met-Hb > 15%].
* Inability to speak English (due to need to administer standardized English-language questionnaire).
* Evidence of anemia.
* History of chronic hemolytic condition, including sickle cell disease.
* Chronic use of anti-migraine medication such as Imitrex or sumatriptan.
* Have a positive screen for glucose-6-phosphate dehydrogenase deficiency at screening.
* Subjects who regularly take the following medications: Allopurinol, PDE-5 inhibitors, sedative tricyclic antidepressants, antihistamines, meperidine and related central nervous system depressants, and nitrates.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Giordano, Ph.D., Study Director — TheraVasc Inc.
Locations (10):
- United States (10):
  - University of Colorado Denver Health Sciences Center, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Mohler ER 3rd, Hiatt WR, Gornik HL, Kevil CG, Quyyumi A, Haynes WG, Annex BH. Sodium nitrite in patients with peripheral artery disease and diabetes mellitus: safety, walking distance and endothelial function. Vasc Med. 2014 Feb;19(1):9-17. doi: 10.1177/1358863X13515043. Epub 2013 Dec 20. PMID 24363302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Started | 18 | 19 | 18
Completed | 15 | 17 | 15
Not Completed | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo twice each day for 11 weeks
- 40 mg Sodium Nitrite: 40 mg dose, BID
  40 mg sodium nitrite: 40 twice each day for 10 weeks followed by a 1 week escalation of 2 times the dose.
- 80 mg Sodium Nitrite: 80 mg dose, BID
  sodium nitrite: 80 mg twice each day for 10 weeks followed by a 1 week escalation of 2 times the dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite | Total
Number analyzed (Participants) | 18 | 19 | 18 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.98) | 65.3 (8.86) | 67.9 (9.99) | 66.0 (9.21)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 4 | 21
  >=65 years | 12 | 8 | 14 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 14
  Male | 13 | 15 | 13 | 41
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 18 | 55

OUTCOME MEASURES:

1. Primary Outcome: Reporting of Adverse Events During 11 Week Treatment Period.
Description: The primary objective of this clinical study is to evaluate the safety and tolerability of multiple doses of twice daily 40mg and 80mg sodium nitrite compared with placebo over a 10 week treatment period. Subjects will be asked to report any adverse events during the trial period, and blood pressure, methemoglobin levels and other blood chemistries will be assessed during the trial period for changes from baseline.
Time Frame: 11 weeks
Measure: Number; unit: participants
Groups:
- Placebo: 0 mg twice each day for 11 weeks.
- 40 mg Sodium Nitrite: 40 mg dose, BID
  sodium nitrite: 40 mg twice each day for 10 weeks followed by a 1 week escalation of 2 times the dose.
- 80 mg Sodium Nitrite: 80 mg dose, BID
  sodium nitrite:80 mg twice each day for 10 weeks followed by a 1 week escalation of 2 times the dose.
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Number analyzed (Participants) | 18 | 19 | 18
participants
  at least 1 AE | 9 | 12 | 14
  SAEs | 2 | 0 | 0

2. Secondary Outcome: Assessment of Changes in Brachial Artery Flow-Mediated Dilation (FMD)at 10 Weeks From Baseline
Description: Demonstrate the pharmacodynamic effect of sodium nitrite on changes in FMD by imaging before investigational product administration and 10 weeks after administration of investigational product but before dose escalation. FMD was measured at baseline and again after 10 weeks of treatment. The value at ten weeks was subtracted from the baseline value. A negative value represents a worsening of FMD while a positive value represents an improvement in FMD.
Time Frame: 10 weeks
Population: Change in flow mediated dilation from baseline to final visit (10 weeks post-treatment)
Measure: Mean (Standard Deviation); unit: percentage from baseline in FMD
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Number analyzed (Participants) | 10 | 15 | 16
percentage from baseline in FMD
  Intent to Treat Population | -2.41 (6.20) | -0.93 (4.58) | 0.06 (3.15)
  Per Protocol Population | -2.69 (6.50) | -0.69 (4.65) | 0.50 (3.28)

3. Secondary Outcome: Assessment of Changes in Walking Distance.
Description: Demonstrate the pharmacodynamic effect of sodium nitrite on changes in functional measures of walking distance. The distance a subject can walk in 6 minutes will be measured prior to the first administration of the investigational product and 10 weeks after taking the investigational product but before the dose escalation. Distance walked in 6 minutes was measured at baseline and again after 10 weeks of treatment. The distance walked at ten weeks was subtracted from the baseline distance walked. A negative value represents a worsening of walking distance while a positive value represents an improvement in walking distance.
Time Frame: 10 weeks
Population: The change in distance walked in 6 minutes at Day 70 compared to baseline.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Number analyzed (Participants) | 17 | 18 | 17
Feet | 7.35 (124.67) | 47.39 (180.46) | -28.82 (259.59)

4. Secondary Outcome: Assessment of Improvement of Quality of Life Using the WIQ (Walking Impairment Questionnaire) and SF-36 Questionnaire.
Description: Demonstrate the pharmacodynamic effect of sodium nitrite on changes in measures of claudication symptoms using Quality of Life questionnaires (WIQ & RAND SF-36). The WIQ is a disease-specific instrument that measures community-based walking. The questionnaire consists of four subscales (pain severity, distance, speed, and stairs). The SF-36 is a set of 36 questions that the subject provides short answers on concerning general health issues that the subject chooses. Questionnaires were administered at baseline and again after 10 weeks of treatment. Scores from the individual sections were summed and divided by the maximal score for the section to obtain a percent score, ranging from 0 (inability to perform task) to 100 (no difficulty). The scores for each section at ten weeks was subtracted from the baseline scores for each section of the questionnaires. A negative represents declining function, a positive value represents improvement over the study period.
Time Frame: 10 weeks
Population: Change in scores on components of quality of life questionnaires at day 70 compared to baseline. The minimum (-100; represents worsening disease) and maximum differences (100, representing complete improvement) from baseline to 10 weeks for the total score of each subsection of the questionnaires are provided.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Number analyzed (Participants) | 17 | 18 | 17
units on a scale
  WIQ: Walking Distance | -1.07 [-14.2 to 45.6] | 2.13 [-70.3 to 63.4] | 5.05 [-66.5 to 61.8]
  WIQ: Walking Speed | 0.00 [-23.9 to 38.0] | 6.52 [-17.4 to 51.5] | 7.07 [-57.6 to 28.3]
  WIQ: Stair Climbing | 0.0 [-41.7 to 45.8] | 12.5 [-25.0 to 58.3] | 0.0 [-37.5 to 45.8]
  SF-36: Physical Functioning | 0.0 [-20.0 to 15.0] | 5.0 [-25.0 to 35.0] | 0.0 [-35.0 to 30.0]
  SF-36: Limitations due to Physcial Health | 25.0 [-75.0 to 50] | 0.0 [-75.0 to 100] | 0.0 [-100.0 to 50]
  SF-36: Limitations due to Emotional Health | 0.0 [-100.0 to 100.0] | 0.00 [-100.0 to 100.0] | 0.0 [-100.0 to 66.7]
  SF-36: Energy/Fatigue | -2.50 [-25.0 to 20.0] | 0.0 [-25.0 to 65.0] | 5.0 [-30.0 to 30.0]
  SF-36: Emotional Well Being | -4.0 [-44.0 to 20.0] | 2.0 [-24.0 to 48.0] | 4.0 [-12.0 to 32.0]
  SF-36: Social Functioning | 0.0 [-25.0 to 12.5] | 0.0 [-25.0 to 62.5] | 0.0 [-37.5 to 50.0]
  SF-36: Pain | 0.0 [-55.0 to 22.5] | 12.5 [-12.5 to 55.0] | 0.0 [-37.5 to 22.5]
  SF-36: General Health | 0.0 [-25.0 to 20.0] | 7.5 [-15.0 to 25.0] | 0.0 [-20.0 to 30.0]

ADVERSE EVENTS:
Groups:
- Placebo: sodium nitrite: 0 mg twice each day for 11 weeks .
Arm/Group | Placebo | 40 mg Sodium Nitrite | 80 mg Sodium Nitrite
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 9/18 | 12/19 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | 40 mg Sodium Nitrite (N=19) | 80 mg Sodium Nitrite (N=18)
Worsening PAD (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | 40 mg Sodium Nitrite (N=19) | 80 mg Sodium Nitrite (N=18)
Headaches and dizziness (General disorders) | 0 (0) | 4 (4) | 8 (8)
GI Disorders (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Infections (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Muscoskeletal and Connective Tissues (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Investigations (Investigations) | 3 (3) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less